CLINICAL TRIAL: NCT00761865
Title: Lateral Ankle Sprain Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low enrollment
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Benedict Digiovanni, Principal Investigator, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23552
Record Dates: First submitted 2008-09-29; First posted 2008-09-30 (Estimated); Results first posted 2015-08-07 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Lateral Ankle Sprain
Keywords: Lateral Ankle Sprin; Air Cast Stirrup Brace; High Tide Fracture Boot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Air Cast Stirrup Brace (Active Comparator): 50 patients will be randomly assigned to receive the Air Cast Stirrup Brace.
  Interventions: Device: Air Cast Stirrup Brace & High Tide Fracture Boot
- High Tide Fracture Boot (Active Comparator): 50 patients will be randomly assigned to the High Tide Fracture Boot.
  Interventions: Device: Air Cast Stirrup Brace & High Tide Fracture Boot

INTERVENTIONS:
Device: Air Cast Stirrup Brace & High Tide Fracture Boot — Subjects will be randomly assigned to one of two treatment braces. All patients will be given instructions to use fracture boot or air cell brace at all times of ambulatory activity until follow-up until 2 week post-strain follow-up.

SUMMARY:
The purpose of this study is to compare the short term treatment outcome measures of the standard of care air cell stirrup brace to that of a high tide fracture boot in patients with lateral ankle sprains.

DETAILED DESCRIPTION:
100 patients with Grade II-III lateral ankle sprains requiring crutches will be invited to participate. Patients will randomly be assigned to be treated with either the Air Cast Stirrup Brace (n=50) or the High Tide Fracture Boot (n=50). All patients will be given instructions to use the fracture boot or air cell brace at all times of ambulatory activity until follow-up and to use NSAIDS as needed. At their 2 week post-sprain follow-up the following outcomes measures will be assessed: Modified Karlsson score (disease specific survey) Pain VAS Patient satisfaction with treatment VAS SMFA (general health measure) Ability to walk without crutches

ELIGIBILITY:
Inclusion Criteria:

* Age 18 & Over
* Lateral Ankle Sprain (Grade II or III) presenting within 48 hours of initial injury without prior treatment

Exclusion Criteria:

* Patients less than 18 years old
* Those not able to give consent
* Women who are pregnant or are expecting to become pregnant
* > 48 hrs from injury at time of presentation
* Prior treatment for injury
* Fracture at time of current ankle injury or previous ankle fracture
* Deltoid ligament injuries
* Other orthopaedic injuries at time of presentation
* Intoxication
* Workman's Compensation injury
* Mental Illness
* Dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benedict DiGiovanni, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Air Cast Stirrup Brace | High Tide Fracture Boot
Started | 16 | 18
Completed | 8 | 11
Not Completed | 8 | 7
Not completed — Lost to Follow-up | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Air Cast Stirrup Brace | High Tide Fracture Boot | Total
Number analyzed (Participants) | 16 | 18 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 18 | 34
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 8 | 13 | 21

OUTCOME MEASURES:

1. Primary Outcome: Modified Karlsson Score
Description: Ankle function score - range 0 to 100. Higher score is better ankle function.
Time Frame: 2 weeks post-sprain
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Air Cast Stirrup Brace | High Tide Fracture Boot
Number analyzed (Participants) | 16 | 18
units on a scale | 67 [33 to 92] | 73 [41 to 95]

2. Secondary Outcome: Patient Satisfaction (Measured on a Visual Analog Scale)
Description: Satisfaction on 0-10 scale with 10 being the best.
Time Frame: 2 weeks post-sprain
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Air Cast Stirrup Brace | High Tide Fracture Boot
Number analyzed (Participants) | 16 | 18
units on a scale | 7 [2 to 9] | 8 [2 to 10]

ADVERSE EVENTS:
Arm/Group | Air Cast Stirrup Brace | High Tide Fracture Boot
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/18
Other Adverse Events (participants affected / at risk) | 0/16 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes